CLINICAL TRIAL: NCT02261740
Title: Program to Overcome Pelvic Pain With Yoga (POPPY) (a.k.a., Development of a Therapeutic Yoga Program for Female Genito-Pelvic Pain)
Brief Title: Program to Overcome Pelvic Pain With Yoga
Acronym: POPPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patty Brisben Foundation For Women's Sexual Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-13946
Record Dates: First submitted 2014-10-01; First posted 2014-10-10 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Pelvic Pain
Keywords: Pelvic Pain; Genital Pain
MeSH Terms: conditions — Pelvic Pain | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga Therapy Group (Experimental): Participants will attend twice-weekly group yoga classes and be instructed to practice yoga at home one additional hour a week, using a written manual.
  Interventions: Behavioral: Yoga Therapy

INTERVENTIONS:
Behavioral: Yoga Therapy — A 90-minute orientation session led by the yoga class instructors, followed by 90-minute group yoga classes twice weekly for 6 weeks. Classes will be led by an experienced instructor. Women will also be taught to avoid any habits that may worsen their genito-pelvic pain (e.g., straining their pelvic floor muscles).
  Participants will also be asked to practice yoga at home an additional hour per week throughout the 6-week yoga therapy program. Participants will be given a detailed written manual to use for home practice.

SUMMARY:
The POPPY Study is a pilot of an Iyengar-based, therapeutic yoga program, used to treat pelvic or genital pain, in up to 16 women. Women aged 21 years and older who report persistent or recurrent pelvic or genital pain for at least 6 months that interferes with sexual activity will be recruited from the San Francisco Bay Area. Those who meet eligibility criteria will take part in a 6-week yoga therapy program designed by an expert yoga panel. Women will attend twice-weekly group classes focusing on Iyengar-based yoga techniques that have been carefully selected for their potential to improve women's genito-pelvic pain and practice yoga at home one additional hour a week.

The investigators will evaluate changes in the severity and impact of women's pain using validated questionnaires and diaries.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 21 years or older who report difficulties with pelvic or genital pain for at least 6 months
2. Report that their chronic pelvic or genital pain has had an adverse effect on their interest in or ability to enjoy sexual activity
3. Report an eligible average daily pain intensity score after completion of a Daily Pain Log for one week prior to baseline
4. Have an established primary care or gynecologic healthcare provider (to facilitate medical follow-up of any health issues detected incidentally in the study or adverse events that develop during the study)
5. Report prior clinical evaluation of their pelvic or genital pain by a health care professional including at least a superficial pelvic exam
6. Willing to refrain from initiating other new clinical treatments that may affect their pelvic or genital pain during the study period (6 weeks)

Exclusion Criteria:

1. Participation in organized yoga classes in the past 1 month, or any prior yoga therapy directed specifically at pelvic or genital pain (regardless of timing)
2. Currently pregnant (by self-report or screening test), pregnant within the past 6 months, planning pregnancy during the study, or unwilling to use contraception (if not postmenopausal) during the study
3. Diagnosed with an alternate cause of pain that is unlikely to respond to yoga and requires another treatment modality, such as pelvic infection or a gynecologic dermatosis
4. Surgery to the vulva, vagina, cervix, or pelvic organs within 6 months of screening, or any prior history of cancer or irradiation to these structures
5. Initiation of or dose escalation of pharmacologic agents that may affect pelvic or genital pain in the past 1 month (e.g., antidepressants, anticonvulsants, anxiolytics)-women on stable dose for >1 month are eligible
6. Use of formal psychological therapies specifically for pelvic or genital pain (e.g., systematic desensitization, sex therapy, cognitive therapy, relaxation therapy) within 1 month of screening
7. Use of formal behavioral therapies for pelvic or genital pain (e.g., pelvic floor rehabilitation or biofeedback performed by a certified healthcare practitioner) within 1 month of screening
8. Unable to walk up a flight of stairs or at least 2 blocks on level ground (i.e., functional capacity < 4 METs), or unable to get up from a supine to a standing position without assistance in <10 seconds
9. Currently involved in a malpractice suit or other litigation specifically related to pelvic or genital pain
10. Participation in another interventional study that might interfere with or confound study procedures, inability to sign an informed consent or fill out questionnaires, or conflict with available yoga class dates

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in severity of pelvic pain after yoga therapy program. | Baseline to 6-Weeks
  Self-reported daily pain severity, as rated by Daily Pain Log (scale from 0-10).

SECONDARY OUTCOMES:
Change in baseline sexual functioning after yoga therapy program. | Baseline, 6-Weeks
  We will use standard questionnaires to assess changes in sexual function.
Change in baseline quality of life after yoga therapy program. | Baseline, 6-Weeks
  We will use standard questionnaires to assess changes in overall quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Huang, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States